## THE IMPACT OF INTRAOPERATIVE LIDOCAINE INFUSION ON POSTOPERATIVE RECOVERY AFTER HYSTEROSCOPY: A RANDOMIZED CONTROLLED TRIAL

## STATISTICAL ANALYSIS PLAN 24<sup>th</sup> DECEMBER 2024

Collected data were analyzed using Statistical Package for Social Sciences version 25.0 (SPSS, IBM Armonk, NY, USA). Kolmogorov-Smirnov test was used to test data distribution. Continuous variables were expressed as mean  $\pm$  standard deviation and categorical variables were presented as frequencies and percentages where appropriate. Student's t-test was used to compare the continuous variables of the study and control groups whereas chi-square test was used to compare the categorical variables of the study and control groups. Two-tailed p values less than 0.05 were accepted as statistically significant.

A post hoc analysis was carried out to make a retrospective power analysis and it was determined that a cohort size of 150 women (75 patients in the study group and 75 patients in the control group) had 87.6 % power to detect a difference at the 0.05 significance level.